CLINICAL TRIAL: NCT00560144
Title: Multiple Ascending Dose (MAD) Study of the IGF-1R Antagonist R1507 Administered as an Intravenous Infusion in Pediatric Patients With Advanced Solid Tumors.
Brief Title: A Multiple Ascending Dose Study of R1507 in Children and Adolescents With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO21200; NCT00557271 (obsolete NCT alias)
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — RG-1507 monoclonal antibody

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: RG1507
- 2 (Experimental)
  Interventions: Drug: RG1507
- 3 (Experimental)
  Interventions: Drug: RG1507

INTERVENTIONS:
Drug: RG1507 — 3mg/kg iv weekly
  Arms: 1
Drug: RG1507 — 9mg/kg iv weekly
  Arms: 2
Drug: RG1507 — Pharmacokinetic-derived dose, <=16mg/kg iv weekly
  Arms: 3

SUMMARY:
This 3 arm study will determine the dose of R1507 which will achieve a mean drug exposure in children and adolescents with advanced solid tumors equivalent to the exposure achieved in adults at the recommended dose of 9mg/kg/week. It will also determine the maximum tolerated dose (if appropriate) and the pharmacokinetic profile of R1507. Groups of patients will be sequentially enrolled in one of up to 3 dose levels (3,9mg/kg or a PK-derived dose, not to exceed 16 mg/kg) of R1507 administered weekly by intravenous infusion.An expanded cohort of patients will be enrolled at the optimal dose/MTD. The anticipated time on study treatment is until disease progression or dose limiting toxicity, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aged 2-17 years of age;
* histologically confirmed solid tumors;
* cancer which has relapsed after, or failed to respond to, curative therapy, or no other potentially curative treatment options available.

Exclusion Criteria:

* treatment with corticosteroids within past 2 weeks;
* current or past use of anti-IGF-1R antibodies;
* current treatment with immunosuppressive agents;
* patients with diabetes mellitus;
* known HIV or hepatitis B or C;
* hypersensitivity to any of the components of R1507 or to monoclonal antibodies.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Serum drug exposure level equivalent to exposure in adults at adult recommended dose. | Throughout study

SECONDARY OUTCOMES:
MTD (AEs, laboratory parameters) | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (6):
  - Tucson, Arizona
  - Denver, Colorado
  - Bethesda, Maryland
  - New York, New York
  - Philadelphia, Pennsylvania
  - Houston, Texas